CLINICAL TRIAL: NCT04412681
Title: Using Precision Medicine for the Prediction and Prevention of Early Pre-eclampsia: A Feasibility Study at Sunnybrook Health Sciences Centre.
Brief Title: Precision Medicine for Prediction & Prevention of Early Pre-eclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: North York General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PEprotocol
Record Dates: First submitted 2020-04-16; First posted 2020-06-02 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PE Enhanced Screening (Experimental): The PE screening program entails the following for all participants:
  * provision of additional demographic and risk factors
  * provision of mean arterial pressure
  * standard nuchal translucency scan as part of their first trimester screening (FTS) with the addition of the measurement of the uterine artery Doppler by a certified sonographer
  * standard blood sample (as part of the FTS)
  * results of the PE screening (in the format of a screening report) will be provided to the study team and participant's healthcare provider
  Interventions: Diagnostic Test: Enhanced PE Screening

INTERVENTIONS:
Diagnostic Test: Enhanced PE Screening — To better identify women at risk for pre-eclampsia during pregnancy.

SUMMARY:
This study aims to evaluate the feasibility of implementing a clinical model for precision screening of early pre-eclampsia into the current prenatal screening service at Sunnybrook Health Sciences Center (SHSC).

DETAILED DESCRIPTION:
Pre-eclampsia (PE) represents a pregnancy-specific systemic disorder that affects 3-8% of all pregnancies. In developed countries PE is considered a major public health problem responsible for severe maternal complications such as coagulopathy, renal and liver failure, stroke, and maternal death (>76,000 maternal death annually).

The traditional approach to screening for preeclampsia endorsed by national guidelines is based on a combination of maternal characteristics along with medical, obstetric and family history.

However, although these methods are simple and easy to perform, maternal factors can only identify less than 35% of all preeclampsia and approximately 40% of preterm-preeclampsia at a false- positive rate of 10%.

More recently, multivariate analysis has been used to develop predictive models for preeclampsia that can be applied as early as 11-13+6 weeks gestation. One such algorithm, developed by the Fetal Medicine Foundation UK(MFM UK), incorporates maternal risk factors, uterine artery doppler, mean arterial pressure, and serum markers of placental function and placental growth factor. The FMFUK algorithm has been shown to predict approximately 75-90% of those women destined to develop preeclampsia prior to 37 and 34 weeks respectively, at a false positive rate of 10%. This algorithm has been validated prospectively in several studies, including the prediction of other placental mediated complications of pregnancy, such as fetal growth restriction and perinatal death.

The new clinical model will include the following additions to the existing first trimester screening for aneuploidy:

* Additional Clinical History
* Blood pressure measurements
* Ultrasound for uterine artery Doppler measurements
* Expanded prenatal screening requisition
* Quality assurance training of ultrasound technicians for the uterine artery doppler measurements
* Fetal Medicine Foundation validated risk calculation algorithm
* Communicate results of the risk calculation algorithm from NYGH to SHSC and participant health care providers.

While the ultimate goal will be to scale up and adapt this new clinical model, this protocol focuses on the feasibility of implementing the new clinical model at a single centre, Sunnybrook Health Sciences Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton pregnancy > 18 years old
2. Not on low dose aspirin
3. Carrying a live fetus with crown rump length (CRL) between 41 and 84mm
4. Able to provide informed consent
5. Having a nuchal translucency ultrasound

Exclusion Criteria:

1. Women with a singleton pregnancy < 18 years old
2. Women currently taking low dose aspirin
3. Women declining a nuchal translucency ultrasound
4. Women unable to provide informed consent
5. Women with a multiple pregnancy
6. Women with a demised fetus or a CRL <41mm and >84mm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Screening Tool | 11.3-13.6 weeks gestation
  Implementation of the screening: To assess the feasibility, the investigators will judge success if the full screening process without deviation is completed for at least 90% of consented participants.

SECONDARY OUTCOMES:
Accuracy of Screening | 11.3-13.6 weeks gestation
  Reproducibility of the FMFUK studies. Planning a recruitment of 1000 participants and anticipating a 10% positive rate, the invetigators expect to follow 100 screen positive and 900 screen negative pregnancies.
Acceptability of Screening Tool to Participants | 11.3-13.6 weeks gestation
  Proportion of acceptance/offer to implementation study. The investigators expect to obtain consent from 80% of pregnant women eligible for the study.
Compliance with low dose ASA for screen positive participants. | 16-36 weeks gestation
  The investigators will assess the rate of initiation and maintenance of low dose ASA ( SHSC standard of care) as measured by phone follow-up at 16,22,26,32 and 36 weeks gestation, (2) follow-up at placental scan visit and (3) follow-up at delivery. Success will defined as 80% compliance.

OTHER OUTCOMES:
Duration of the assessment | 11.3-13.6 weeks gestation
  The investigators will assess the duration (in minute) required for completing data questionnaire, measuring arterial blood pressure and uterine artery Doppler
Turnaround time from assessment to results | 11.3-16 weeks gestation
  The investigators will measure the turnaround time (in business day) from screening requisition reaching laboratory to report issued to SHSC via fax
Participant Satisfaction | 11.3-40 weeks gestation
  The investigators will assess participant satisfaction with screening and care through a satisfaction survey with a 10 score scale where 1 is very unsatisfied and 10 is very satified

CONTACTS AND LOCATIONS:
Overall Officials: Ronzoni, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Health Sciences center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Wright D, Syngelaki A, Akolekar R, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal characteristics and medical history. Am J Obstet Gynecol. 2015 Jul;213(1):62.e1-62.e10. doi: 10.1016/j.ajog.2015.02.018. Epub 2015 Feb 25. PMID 25724400
- [Background] O'Gorman N, Wright D, Poon LC, Rolnik DL, Syngelaki A, de Alvarado M, Carbone IF, Dutemeyer V, Fiolna M, Frick A, Karagiotis N, Mastrodima S, de Paco Matallana C, Papaioannou G, Pazos A, Plasencia W, Nicolaides KH. Multicenter screening for pre-eclampsia by maternal factors and biomarkers at 11-13 weeks' gestation: comparison with NICE guidelines and ACOG recommendations. Ultrasound Obstet Gynecol. 2017 Jun;49(6):756-760. doi: 10.1002/uog.17455. PMID 28295782
- [Background] Park FJ, Leung CH, Poon LC, Williams PF, Rothwell SJ, Hyett JA. Clinical evaluation of a first trimester algorithm predicting the risk of hypertensive disease of pregnancy. Aust N Z J Obstet Gynaecol. 2013 Dec;53(6):532-9. doi: 10.1111/ajo.12126. Epub 2013 Aug 6. PMID 23919594
- [Background] Mosimann B, Pfiffner C, Amylidi-Mohr S, Risch L, Surbek D, Raio L. First trimester combined screening for preeclampsia and small for gestational age - a single centre experience and validation of the FMF screening algorithm. Swiss Med Wkly. 2017 Aug 25;147:w14498. doi: 10.4414/smw.2017.14498. eCollection 2017. PMID 28871576
- [Background] O'Gorman N, Wright D, Poon LC, Rolnik DL, Syngelaki A, Wright A, Akolekar R, Cicero S, Janga D, Jani J, Molina FS, de Paco Matallana C, Papantoniou N, Persico N, Plasencia W, Singh M, Nicolaides KH. Accuracy of competing-risks model in screening for pre-eclampsia by maternal factors and biomarkers at 11-13 weeks' gestation. Ultrasound Obstet Gynecol. 2017 Jun;49(6):751-755. doi: 10.1002/uog.17399. Epub 2017 May 14. PMID 28067011
- [Background] Ananth CV, Keyes KM, Wapner RJ. Pre-eclampsia rates in the United States, 1980-2010: age-period-cohort analysis. BMJ. 2013 Nov 7;347:f6564. doi: 10.1136/bmj.f6564. PMID 24201165
- [Derived] Ronzoni S, Rashid S, Santoro A, Mei-Dan E, Barrett J, Okun N, Huang T. Preterm preeclampsia screening and prevention: a comprehensive approach to implementation in a real-world setting. BMC Pregnancy Childbirth. 2025 Jan 15;25(1):32. doi: 10.1186/s12884-025-07154-6. PMID 39815166